CLINICAL TRIAL: NCT03692819
Title: Effect of Antibiotic and Probiotic Therapies in the Adjuvant Treatment of Chronic Periodontitis: Randomized Controlled Clinical Trial.
Brief Title: Antibiotic and Probiotic Therapies in the Adjuvant Treatment of the Chronic Periodontitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Maria Aparecida Neves Jardini, Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Probioticos e Antibióticos
Record Dates: First submitted 2018-09-06; First posted 2018-10-02 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Chronic Periodontitis Complex
Keywords: Chronic Periodontitis; Periodontal Debridement; Antibiotics; Probiotics
MeSH Terms: conditions — Chronic Periodontitis | interventions — Periodontal Debridement; Amoxicillin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective double-blind randomized controlled clinical study with a 90-days follow-up.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition to concealment of randomization, the investigator responsible for the procedures of periodontal therapy (periodontal debridement) and the researcher responsible for the measurements will not know which treatment each group will receive, characterizing the blindness of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Active Comparator): Periodontal debridement treatment will be performed in a single session after the therapy will be administered the Placebo Oral Tablet twice a day for 21 days.
  Interventions: Drug: Placebo Oral Tablet
- Metronidazole and Amoxicillin (Experimental): Periodontal debridement treatment in a single session Metronidazole 400mg + Amoxicillin 500mg every 8 hours for 7 days.
  Interventions: Drug: Amoxicillin 500 Mg
- Lactobacillus reuteri (Experimental): Periodontal debridement treatment in a single session Lactobacillus reuteri Oral Drops twice a day for 21 days.
  Interventions: Drug: Lactobacillus reuteri Oral Drops

INTERVENTIONS:
Drug: Placebo Oral Tablet — Non-surgical periodontal treatment will be performed by means of periodontal debridement in a single session.
  Other Names: Periodontal debridement
  Arms: placebo
Drug: Amoxicillin 500 Mg — Non-surgical periodontal treatment will be performed by means of periodontal debridement in a single session after the therapy will be administered the antibiotic (Metronidazole 400mg + Amoxicillin 500mg) every 8 hours for 7 days
  Other Names: Metronidazole Oral
  Arms: Metronidazole and Amoxicillin
Drug: Lactobacillus reuteri Oral Drops — Non-surgical periodontal treatment will be performed by means of periodontal debridement in a single session after the therapy will be administered the probiotic (Lactobacillus reuteri oral drops ) twice a day for 21 days.
  Other Names: Prodentis
  Arms: Lactobacillus reuteri

SUMMARY:
Currently, with the increase of bacterial resistance to antibiotics associated with its side effects, it is necessary to find other adjuncts to combat the disease that are an alternative to the use of antibiotics. The use of probiotics has been proposed in the literature as an adjunct therapy for the treatment of periodontal diseases, however, few controlled and randomized clinical studies have been performed. The objective of this double-blind randomized controlled trial will be to evaluate the response of clinical and microbiological periodontal parameters to the comparison of two different adjuvant therapies (antibiotic and probiotic) for the treatment of stages II and III grade B periodontitis.

DETAILED DESCRIPTION:
Currently, with the increase of bacterial resistance to antibiotics associated with its side effects, it is necessary to find other adjuncts to combat the disease that are an alternative to the use of antibiotics. The use of probiotics has been proposed in the literature as an adjunct therapy for the treatment of periodontal diseases, however, few controlled and randomized clinical studies have been performed. The objective of this double-blind randomized controlled trial will be to evaluate the response of clinical and immunological periodontal parameters to the comparison of two different adjuvant therapies (antibiotic and probiotic) for the treatment of stages II and III grade B periodontitis. Patients will be randomized into 3 groups: Group 1 (n=15): periodontal debridement, Group 2 (n=15): periodontal debridement associated with antibiotic (Metronidazole 400 mg + Amoxicillin 500mg) and Group 3 (n=15): periodontal debridement associated with probiotic (Lactobacillus reuteri). Clinical (plaque index, gingival index, probing depth, gingival recession, relative clinical attachment level and periodontal inflamed surface area (PISA) index) and immunological data obtained before and after periodontal therapy (baseline, 30 and 90) will be consolidated and made available on average ± standard deviation and normality tested using the Shapiro-Wilk test. For statistical analysis, the software BioEstat 5.0 (Belém, PA, Brazil) will be used, with p-value < 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 35 and 50 years of age;
* Be diagnosed with generalized chronic periodontitis: present a loss of interproximal clinical insertion> 3 mm in 2 nonadjacent teeth and loss of interproximal clinical insertion ≥5 mm, in 30% or more of the teeth present;
* Present at least 16 teeth;
* Present good systemic health;
* Agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Patients with systemic problems (cardiovascular changes, blood dyscrasias, immunodeficiency, among others), which do not indicate the periodontal procedure;
* Have undergone periodontal treatment in the last twelve months;
* Have used antibiotics and/or anti-inflammatories for the past six months;
* Smoking patients;
* Pregnancy or Lactation;
* Chronic use of medications that may alter the response of periodontal tissues.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Probing Depth change | Baseline, 30 and 90 days
  The change in the probing depth will be measure in millimeters before and after the treatment.

SECONDARY OUTCOMES:
Plaque Index | Baseline, 30 and 90 days
  Number of teeth affected before and after periodontal treatment.
Gingival Index | Baseline, 30 and 90 days
  Number of teeth affected before and after the treatment.
Gingival Recession | Baseline, 30 and 90 days
  Evaluated in milimeters before and after the treatment.
Clinical Attachment Level | Baseline, 30 and 90 days
  Evaluated in milimeters before and after the treatment.
Periodontal Inflamed Surface Area (PISA) | Baseline, 30 and 90 days
  Is calculated from data collected on probing the periodontal pocket and are placed in a table which gives the value of the periodontal inflamed surface area.
Microbiological Parameters | Baseline, 30 and 90 days
  crevicular fluid samples will be analyzed by PCR (real time PCR) for detection and quantification of: Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola and Lactobacillus reuteri.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jardini, PhD, Study Director — Universidade Estadual Paulista Julio de Mesquita Filho
Locations (1):
- Maria Jardini, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No